CLINICAL TRIAL: NCT04606719
Title: Healing Potentiality Of Blood Clot, S-PRF and A-PRF As Scaffold In Treatment Of Non-Vital Mature Single Rooted Teeth With Chronic Peri-Apical Periodontitis Following Regenerative Endodontic Therapy (Randomized Clinical Trial)
Brief Title: Healing Potentiality Of Blood Clot S-PRF and A-PRF in the Treatment Of Necrotic Mature Single-Rooted Teeth With Chronic Peri-Apical Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Badawy Darwish, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENDO 5-6-1
Record Dates: First submitted 2020-10-25; First posted 2020-10-28 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Necrotic Pulp
Keywords: Regeneration . Necrotic . Mature teeth . Blood clot . PRF
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Blood Clot (Other): It is induced through apical foramen by penetrating the periapical area by stainless steel file size 30 to fill the root canal system by growth factors also to be considered as scaffold
  Interventions: Procedure: Advanced Platelet Rich fibrin
- Standard PRF (Active Comparator): Standard Platelet-rich fibrin will be prepared by drawing 5 mL of venous blood from the patient in dried glass test tube and immediately centrifuging it at 3000 rpm for 10 min. After centrifugation, three layers will formed in the test tube-base layer of RBCs, top layer of a-cellular plasma, and a PRF clot in the middle. This clot will then pressed between two gauze pieces to form a membrane.
  Interventions: Procedure: Advanced Platelet Rich fibrin
- Advanced PRF (Experimental): A-PRF by drawing 5 mL of venous blood from the patient in dried glass test tube and immediately centrifuging it at 1500 rpm for 14 minutes
  Interventions: Procedure: Advanced Platelet Rich fibrin

INTERVENTIONS:
Procedure: Advanced Platelet Rich fibrin — Preparing of A-PRF by drawing 5 mL of venous blood from the patient in dried glass test tube and immediately centrifuging it at 1500 rpm for 14 minutes

SUMMARY:
Earlier, it was believed that successful regeneration cannot be achieved once tooth has become infected. However, recent studies suggest that regenerative endodontics may in fact be possible in teeth with pulpal necrosis and periapical pathology.

The primary goal in regenerative procedure is to eliminate clinical symptoms and resolve apical periodontitis. The blood clot acts as a scaffold, and the growth factors inside recruit stem cells, most likely from periapical papilla. But unfortunately, the erythrocytes in the clot of the blood column undergo necrosis, affecting its properties so the blood column is augmented by the use of different types of scaffolds.

Platelet-rich fibrin is classified into four types (Standard PRF, Injectable PRF, Advanced PRF and Concentrated Growth Factor CGF) according to speed and time of centrifuge with the overall aim to increase the number of platelets and leucocytes

ELIGIBILITY:
Inclusion Criteria:

* Medically free patients who accept to participate in the study.
* Age between 18-35 years old with no sex predilection.
* Patients with good oral hygiene.
* Patients with necrotic pulp in mandibular & maxillary single rooted permanent teeth with mature apex that Symptomatic or Asymptomatic , Doesn't respond positively with the electric pulp tester ,Associated with or without swelling /sinus tract, Has radiographic evidence of periapical radiolucency, Has a straight, non-curved root, Teeth with normal occlusal contact with the opposing teeth.

Exclusion Criteria:

* Illiterate patient because they can't estimate the pain level on the pain scale (NRS).
* Patients with systemic diseases or on systemic corticosteroids therapy because they have impaired healing and higher incidence of pain.
* Pregnant women to avoid radiation exposure during the treatment which may be hazardous to the fetus and breasts from dental X-ray examinations shields.
* Patients that have allergy to ciprofloxacin or metronidazole to avoid any allergic reaction after placement of bi-antibiotic paste as intra-canal medication.
* Patients reporting bruxism or clenching because this induce more pressure on teeth and may initiate the post-operative pain in the treated tooth which is already have peri-apical inflammation
* Teeth that, Have vertical root fracture, coronal perforation, and calcification, Are indicated for retreatment because they have lower success rate , Have pocket depth greater than 5mm,Need periodontal therapy , Non restorable , Hopeless tooth, patients that have T.M.J disorder

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
healing Rate | follow up to 6 months
  standardized digital radiograph

SECONDARY OUTCOMES:
Postoperative pain: NRS | up to one year
  using neumerical rationg scale NRS . from zero to 10 . zero = no pain 1 to 3 = mild 4-6 = moderate 7-10 = severe
sensitivty | 6 months to one year
  using sensitivity tests

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Derived] Darwish OB, Aziz SMA, Sadek HS. Healing potentiality of blood clot, S-PRF and A-PRF as scaffold in treatment of non-vital mature single rooted teeth with chronic peri-apical periodontitis following regenerative endodontic therapy: randomized clinical trial. BMC Oral Health. 2025 Jan 9;25(1):50. doi: 10.1186/s12903-024-05378-0. PMID 39789544